CLINICAL TRIAL: NCT02299648
Title: The Screening Protocol for The VIKTORY Trial- Targeted Agent eValuation in gastrIc Cancer basKeT KORea studY: SMC-AZ GC Basket Trial Screening Protocol
Brief Title: The Screening Protocol for The VIKTORY Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014-04-119-009
Record Dates: First submitted 2014-10-16; First posted 2014-11-24 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): molecular profiling, patient derived cells
  Interventions: Other: Molecular profiling

INTERVENTIONS:
Other: Molecular profiling — molecular profiling, patient derived cells, fresh or FFPE

SUMMARY:
This protocol is a screening protocol only. No drug intervention study will be included in this protocol. However, based on the molecular profiling, patients may be eligible for targeted agents. However, the molecular profiling doesn't guarantee the enrollment onto the clinical trial. Currently, the available drugs are AKT inhibitor, MEK inhibitor, Wee1 inhibitor, MET inhibitor. ATR inhibitor and other agents may be available in the context of clinical trials depending on the availability.

DETAILED DESCRIPTION:
To screen metastatic GC patients who failed or progressed on first-line chemotherapy. Patients will undergo biopsy of their tumor and will be analyzed using cancer panel/nanostring CNV and immunohistochemistry. This protocol is a screening protocol and informed consent form will be obtained again according to the biomarker profiled on this protocol if eligible. Informed consent will be obtained from patients with gastric adenocarcinoma and analysis of fresh tissue or archival FFPE at Samsung Medical Center will be performed. Patients who have prior to or completed or during the first-line chemotherapy (fluoropyramidine/platinum-based) will be eligible for screening.

After the analysis, pathologic and molecular biologic verification process about validity of the result will proceed. The biopsies will be performed before or after or during first-line treatment for molecular analysis. The patients who are screened through this protocol will undergo baseline biopsy before or after or during first-line therapy.

Study Objectives

1. Primary Objective: To screen metastatic GC patients who failed or progressed on first-line chemotherapy. Patients will undergo biopsy of their tumor and will be analyzed using cancer panel/nanostring CNV and immunohistochemistry.
2. Secondary Objective

Planned subgroup analyses:

1. OS (biomarker negative vs biomarker postivie metastatic GC patients)
2. PFS (biomarker negative vs biomarker postivie metastatic GC patients)
3. OS/PFS (EBV negative vs positive metastatic GC patients)

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Metastatic or recurrent esophageal, gastroesophageal or gastric adenocarcinoma
* Progressed and/or completed one platinum/fluoropyrimidine-based cytotoxic chemotherapy regimen (any adjuvant treatment will not be considered as one palliative regimen): patients who have prior to or completed or during first-line chemotherapy will be eligible for screening.
* Tissue specimens: surgical specimens, endoscopic biopsies, colono/sigmoidoscopic biopsies, liver biopsies, lymph node biopsies, malignant cells isolated from ascites/pleural effusion/pericardial effusion/other malignancy related body fluids with sufficient number of malignant cells for DNA/RNA extractions will be allowed.
* Age ≥ 20 years 5) ECOG performance status 0-1 6) Written informed consent - Life expectancy ≥ 3 months
* Patients with available archival tissues for molecular analysis or patients who agreed with biopsy for molecular analysis (however, fresh frozen tissue will be considered first)

Exclusion Criteria:

* Prior history of taxane treatment as palliative chemotherapy
* Uncontrolled systemic illness and infection
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2014-07-25 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
molecular screening ( biopsy of their tumor and will be analyzed using cancer panel/nanostring CNV and immunohistochemistry) | from data of start of targeted tretment oriented by molecular screening until the date of first progression or date of death form any cause, whichever came first, assessed up to 1 year
  To screen metastatic GC patients who failed or progressed on first-line chemotherapy. Patients will undergo biopsy of their tumor and will be analyzed using cancer panel/nanostring CNV and immunohistochemistry.

SECONDARY OUTCOMES:
OS | 1years
  OS (biomarker negative vs biomarker postivie metastatic GC patients)
PFS | 1years
  PFS (biomarker negative vs biomarker postivie metastatic GC patients)
OS/PFS | 1years
  OS/PFS (EBV negative vs positive metastatic GC patients)

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, MD, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical center, Seoul
  - Samsung Medical Center, Seoul